CLINICAL TRIAL: NCT00928538
Title: Effectiveness of Home Based Distribution of Hormonal Contraceptives for Women at Risk for Unintended Pregnancy
Brief Title: Nurse Family Partnership (NFP) Contraceptive Study
Acronym: NFP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Colorado, Denver (Other); Clark County Department of Public Health (Unknown); Thurston County Department of Public Health and Social Services (Unknown); Public Health - Seattle and King County (Other Government)
Responsible Party: Principal Investigator, Alan Melnick, Adjunct Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 832
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy; Effective Contraceptive Use; Family Planning
Keywords: Female Contraception; Home Visits; CONTRACEPTIVE AGENTS; CONTRACEPTIVE DEVICES

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual NFP Care (No Intervention): Usual NFP care includes pregnancy planning and contraceptive advice during nurse home visits, with the prescription and dispensing of contraceptives provided through the women's primary care settings.
- Enhanced NFP Care (Experimental): Enhanced NFP intervention includes usual NFP care plus the intervention that includes contraceptive administration and distribution in the home
  Interventions: Other: Enhanced NFP Care

INTERVENTIONS:
Other: Enhanced NFP Care — Usual NFP care plus the enhanced care that includes contraceptive administration and distribution during nurse home visits. Participants will have a choice of combined hormonal contraception (oral, patches or vaginal rings)or progestin-only contraception (oral or depomedroxyprogesterone acetate injections.
  Arms: Enhanced NFP Care

SUMMARY:
The purpose of this study is to determine whether nurses can help at-risk women reduce the incidence of unintended pregnancy by providing them access to hormonal contraceptives in their homes.

DETAILED DESCRIPTION:
The investigators intend to accomplish this goal by strengthening the family planning component of a well-known, effective, home-based intervention, the Nurse Family Partnership (NFP), by enhancing the nurses' access to contraceptive supplies. The investigators believe that proposed modification to the intervention, giving the nurses the ability to deliver hormonal contraception in the home, will enable the nurses to bring about greater change in the reproductive health behavior of women at-risk for unintended pregnancy. Ultimately, the investigators believe this will increase the impact the NFP has had on conception rates during the first two postpartum years.

Participants will be enrolled through the Nurse Family Partnership program in the Public Health Departments in Seattle/King County, Thurston County and Clark County, Washington. The NFP program provides home visits for women anticipating a first birth. Inclusion criteria for participation include English or Spanish speaking (or both), enrolled in the NFP program, pregnant and anticipating a first birth, and 32 weeks or less gestation. NFP nurses will obtain written consent for the study as well as consent for family planning services.

The study will be a randomized clinical trial. After consent and enrollment in the study, we will randomize participants to receive either the usual NFP intervention or the enhanced NFP intervention that includes contraceptive administration and distribution. The usual NFP intervention includes interventions focused on pregnancy planning and contraceptive advice, with the prescription and dispensing of contraceptives provided through the women's primary care settings. The primary difference between routine NFP care and the enhanced intervention is the administration and distribution of hormonal contraception in the home with one exception. Because it is part of the usual intervention, when requested, NFP nurses will provide emergency contraceptives for participants in both arms of the study. Each participant assigned to the enhanced intervention will receive the routine NFP family planning counseling beginning during pregnancy, including information on available contraceptives. The nurse will also counsel participants on when to begin using contraceptives post-partum. Following delivery, the nurse will take a history to determine whether there are any contraindications to oral contraceptives, the contraceptive patch, the contraceptive vaginal ring or the depomedroxyprogesterone shot. The nurse will follow study protocols, approved by the Clark County, Thurston County and Seattle/King County Public Health Departments, when taking the history, and if necessary, obtain a urine pregnancy test. The nurse will obtain written consent for family planning services before providing contraceptives. The written consent form is similar to consent forms used in clinic settings. The nurse will continue to provide family planning counseling, including counseling on sexually transmitted infection (STI) prevention and cervical cancer screening, and a supply of condoms. The nurse will also offer a choice of a three-month supply of combination oral contraceptives, progestin-only oral contraceptives, contraceptive patches, the contraceptive vaginal ring or a depomedroxyprogesterone injection at no cost to the participant. Depending on the contraceptive method chosen, the nurse will provide education, counseling, and obtain written request and consent forms for the specific method. All written materials will be available in English and Spanish. Monolingual Spanish-speaking patients will receive services from Spanish speaking NFP nurses. The nurses will follow guidelines and standing orders developed by Dr. Gipson, the Co-Investigator for the study, subject to approval by the county Health Officer, when providing oral contraceptives, contraceptive patches, or the contraceptive vaginal ring or when administering the depomedroxyprogesterone shot. For women currently breastfeeding, the nurse will recommend and provide progestin-only oral contraceptives or administer the depomedroxyprogesterone shot. During frequent home visits, the NFP nurse will continue to counsel the participants while providing additional three to twelve-month supplies of contraceptives or administering the depomedroxyprogesterone injections for up to two years after delivery. By phone or through subsequent visits, the nurse will address any adverse reactions or other participant concerns and will provide refills or an alternative hormonal method as necessary.

For both groups (usual NFP care and enhanced intervention), the Research Associates (RAs) will gather data related to gaps in contraceptive coverage and repeat pregnancy every three months beginning six months after delivery (except at 12 months and two years postpartum). In addition, RAs will conduct phone surveys following enrollment and again at 3 months, 12 months and 24 months post delivery. The surveys will address factors that influence the rate and timing of subsequent pregnancy, including pregnancy intendedness, utilization of reproductive health services, perceived barriers to contraceptive use, satisfaction with birth control methods, and self-efficacy related to contraceptive use.

Aim 1 is to determine whether fewer participants in the enhanced intervention group experience more than a one month gap in effective contraceptive use (defined as methods with which < 10% of women experience an accidental pregnancy during a year of typical use) compared to participants in the usual care group. The investigators will answer this by comparing the incidence of gaps that occur in the twenty-four months after delivery using survival analysis methods. Aim 2 is to examine whether fewer participants in the enhanced intervention group experience a second pregnancy compared to participants in the usual care group. The methodology for Aim 2 will be the same as for Aim 1, with analysis based on incidence of second pregnancy rather than gap in effective contraceptive use. Aim 3 will be to explore how pregnancy intendedness modifies the outcomes in Aim 1 and Aim 2, using the same methodology as aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking (or both)
* Enrolled in the NFP (Nurse Family Partnership) program
* 32 weeks or less gestation.

Exclusion Criteria:

* Not enrolled in the NFP program
* More than 32 weeks gestation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 344 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
One month gaps in effective contraceptive use (defined as methods with which < 10% of women experience an accidental pregnancy during a year of typical use) | Every three months after delivery for two years

SECONDARY OUTCOMES:
Unintended pregnancy | Every three months after delivery for two years

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Melnick, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Thurston County Public Health, Olympia, Washington
  - Seattle - King County Public Health, Seattle, Washington
  - Clark County Public Health, Vancouver, Washington

REFERENCES:
- [Background] Melnick AL, Rdesinski RE, Creach ED, Choi D, Harvey SM. The influence of nurse home visits, including provision of 3 months of contraceptives and contraceptive counseling, on perceived barriers to contraceptive use and contraceptive use self-efficacy. Womens Health Issues. 2008 Nov-Dec;18(6):471-81. doi: 10.1016/j.whi.2008.07.011. Epub 2008 Oct 15. PMID 18926726
- [Background] Rdesinski RE, Melnick AL, Creach ED, Cozzens J, Carney PA. The costs of recruitment and retention of women from community-based programs into a randomized controlled contraceptive study. J Health Care Poor Underserved. 2008 May;19(2):639-51. doi: 10.1353/hpu.0.0016. PMID 18469433